CLINICAL TRIAL: NCT06095934
Title: Exploration of the Efficacy and Safety of Anti-PD-1 Monoclonal Antibody Combined With Neoantigen Peptide Vaccine and Chemotherapy in the Treatment of Advanced NSCLC Progressed After EGFR-TKI Treatment
Brief Title: Efficacy and Safety of Neoantigen Peptide Vaccine in the Treatment of Advanced NSCLC Progressed After EGFR-TKI Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yang Yang, Principal Investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEOVAC-BGB-C
Record Dates: First submitted 2023-09-07; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: NSCLC; EGFR Gene Mutation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluate the efficacy and safety of neo-antigen peptide vaccine in the treatment of advanced NSCLC (Experimental)
  Interventions: Other: neo-antigen vaccine

INTERVENTIONS:
Other: neo-antigen vaccine — anti-PD-1 monoclonal antibody combined with neoantigen peptide vaccine and chemotherapy

SUMMARY:
To evaluate the efficacy (ORR) and safety of anti PD-1 monoclonal antibody combined with neoantigen peptide vaccine and chemotherapy in the treatment of advanced NSCLC progressed after EGFR-TKI treatment and to provide new treatment methods for EGFR-TKI resistant patients.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily joined this study and signed an informed consent form;
2. ≥ 18 years old, both male and female;
3. Pathologically confirmed IIIB-IV stage NSCLC, with at least one measurable lesion that has not undergone local treatment (according to RECIST v1.1, the length of the measurable lesion on spiral CT or MRI scans is ≥ 10 mm or the short diameter of the enlarged lymph node is ≥ 15 mm);
4. Metastatic advanced EGFR mutated lung cancer confirmed by histology or cytology, with EGFR-TKI monotherapy or EGFR-TKI combined anti angiogenic therapy failing;
5. Patients who have received first-line chemotherapy in the past can be included in the inclusion criteria;
6. ECOG score: 0-2;
7. Expected survival time ≥ 12 weeks;
8. The functions of important organs meet the following requirements:Absolute neutrophil count ≥ 1.5 × 109/L;Absolute lymphocyte count ≥ 0.8 × 109/L;Platelets ≥ 80 × 109/L;Hemoglobin ≥ 90g/L;Bilirubin ≤ 1.5 × ULN (within 7 days before the first medication);ALT and AST ≤ 1.5 × ULN (within 7 days before the first medication); Serum creatinine ≤ 1.5 × ULN;
9. Thyroid stimulating hormone (TSH) ≤ 1 × ULN (if abnormal, FT3 and FT4 levels should be examined simultaneously, and if FT3 and FT4 levels are normal, they can be included in the group level);
10. For female patients of childbearing age, effective methods of contraception should be used during the trial period and within 3 months after the last administration of treatment medication;
11. Agree to provide blood samples and histological specimens.

Exclusion Criteria:

1. The patient has any active autoimmune disease or a history of autoimmune disease;
2. The patient is currently using immunosuppressive agents or systemic hormone therapy to achieve immunosuppressive effects (dosage>10mg/day of prednisone or other therapeutic hormones) ;
3. The patient experienced severe allergic reactions to other monoclonal antibodies;
4. Suffering from hypertension and unable to achieve good control through antihypertensive medication treatment (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥ 90mmHg);
5. There are clinical symptoms or diseases of the heart that cannot be well controlled, such as:NYHA grade 2 or above heart failure;Unstable angina pectoris; Have experienced myocardial infarction within 1 year;Clinically significant supraventricular or ventricular arrhythmias require treatment or intervention; QTc>450ms (male); QTc>470ms (female);
6. Abnormal coagulation function (INR>2.0, PT>16s), with bleeding tendency or undergoing thrombolysis or anticoagulation treatment, allowing prophylactic use of low-dose aspirin and low molecular weight heparin;
7. Received previous anti-tumor immunotherapy and anti-tumor vaccine treatment;
8. The patient has active infection, unexplained fever ≥ 38.5 ° C within 7 days before medication, or baseline white blood cell count>15 × 109/L; Those who may have purulent or chronic infections, and the wound persists without healing;
9. Patients who have experienced bone metastasis have received palliative radiotherapy in areas greater than 5% of the bone marrow area within the 4 weeks prior to participating in this study;
10. The patient has previously received anti PD-1, anti PD-L1, and anti PD-L2 treatment;
11. Those who are known to be allergic to the components of recombinant humanized anti-PD-1 monoclonal antibody drugs and vaccines;
12. Pregnant or lactating women, or female patients with fertility who have not taken contraceptive measures;
13. Other malignant tumors (excluding basal cell or squamous cell carcinoma, superficial bladder cancer cancer, cervical carcinoma in situ or breast cancer) in the past 5 years;
14. Patients who participate in other clinical trials at the same time;
15. HIV positive; HCV positive; Uncontrolled active hepatitis B;
16. Those who have received live vaccination within 4 weeks before the start of treatment;
17. Patients with a history of asymptomatic brain metastasis who meet all the following conditions can be selected:During screening, brain imaging showed no evidence of immediate progression.There is currently no need to use glucocorticoids to treat brain metastases, and stable doses of anticonvulsants are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | three years
  Exploration of the efficacy of anti-PD-1 monoclonal antibody combined with neoantigen peptide vaccine and chemotherapy in the treatment of advanced NSCLC with previous EGFR-TKI treatment failure

SECONDARY OUTCOMES:
PFS | three years
  Observe and evaluate the progression free survival (PFS), overal survival(OS) of advanced NSCLC patients who have failed previous EGFR-TKI treatment with anti-PD-1 monoclonal antibody combined with neoantigen peptide vaccine and chemotherapy;
OS | three years
  Observe and evaluate the overal survival(OS) of advanced NSCLC patients who have failed previous EGFR-TKI treatment with anti-PD-1 monoclonal antibody combined with neoantigen peptide vaccine and chemotherapy;

CONTACTS AND LOCATIONS:
Locations (1):
- The Comprehensive Cancer Centre of Nanjing Drum Tower Hospital, Medical School of Nanjing University & Clinical Center Institute of Nanjing University, Nanjing, China, Nanjing, China

IPD SHARING:
Plan to Share IPD: No